CLINICAL TRIAL: NCT01797315
Title: Prevention of Skin Cancer in High Risk Patients After Conversion to a Sirolimus-based Immunosuppressive Protocol
Acronym: PROSKIN
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: no adequate recruitment
Sponsor: University Hospital of Berlin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROSKIN 01
Record Dates: First submitted 2013-02-15; First posted 2013-02-22 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2013-02

CONDITIONS: Renal Transplant Patients at High-risk for Skin Cancer
MeSH Terms: interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sirolimus (Active Comparator): Patients who meet all inclusion criteria will be included into the study and randomised. If converted to Sirolimus (SRL), patients will take SRL according to the investigator's instructions and medication label, once daily preferably 4 hours after calcineurin-inhibitor medication or in case without calcineurin-inhibitor co-medication in the morning. The dose of SRL will be correlated to the former immunosuppressive therapy according to the study's conversion protocol.
  Interventions: Drug: Sirolimus
- Standard therapy (No Intervention): Patients who will not receive SRL stay on their previous immunosuppressive therapy including one or more of the following drugs: azathioprine, cyclosporine, tacrolimus, mycophenolate-sodium and steroids.

INTERVENTIONS:
Drug: Sirolimus
  Other Names: Rapamune®
  Arms: Sirolimus

SUMMARY:
Transplant recipients have a high risk to develop skin malignancies. This effect depends on the one hand on the immunosuppressive drugs themselves and relates on the other hand on the dosage. Based on the encouraging results of previous, retrospective studies on patients treated with Sirolimus (SRL), these patients should be switched to an immunosuppressive regime including SRL, decreasing the dosage of calcineurin-inhibitors or converting from former immunosuppression. A conversion to a SRL-based therapy is effective in immunosuppression and safe regarding graft and patient survival.

This study was designed to assess whether a switch to a SRL-immunosuppressive therapy decreases the incidence/reoccurrence of skin neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of renal allograft with current actinic keratosis I or II or successfully treated actinic keratosis III (inclusion possible immediately after completed wound healing from surgical excision), invasive squamous cell carcinoma (SCC), basal cell carcinoma
* age 18 years and older
* minimum period of 6 month after renal transplantation
* stable renal function and a calculated creatinine clearance of at least 40 ml/min
* written informed consent
* proteinuria ≤ 800 mg/d at time of enrolment
* successfully treated solid tumor (no recurrence or metastasis in the last 2 years)

Exclusion Criteria:

* Current Sirolimus- or Everolimus- intake
* Instable graft function (creatinine clearance < 40 ml/min)
* Graft rejection within the 3 previous months
* Proteinuria > 800 mg/d
* Non-controlled hyperlipidemia (Cholesterol >7,8 mmol/l (300 mg/dl), Triglycerides > 4 mmol/l (350 mg/dl)
* Leucopenia < 2500/nl
* Thrombocytopenia < 90/nl
* Pregnancy or breastfeeding
* Women of childbearing age without highly effective contraception
* Known allergy to macrolides
* Current participation in other studies
* Refusal to sign informed consent form
* Neoplasm other than defined as inclusion criteria
* All contraindications to SRL (see package insert, appendix)
* Persons who are detained officially or legally to an official institute
* Acute infections (mycotic, viral or bacterial)
* Current intake of other substances with known nephrotoxicity
* Severe liver dysfunction
* Current intake of CY3A4-inhibitors (e.g. ketoconazole, voriconazole, itraconazole, telithromycin or clarithromycin) or CY3A4-inductors (rifampicin, rifabutin)
* sucrose-isomaltase deficiency, fructose intolerance, glucose-galactose intolerance
* azathioprine: known allergy to azathioprine or 6-mercaptopurine, severe bone marrow dysfunction, pancreatitis, vaccination with live vaccine
* tacrolimus: known allergy to tacrolimus
* mycophenolatmofetil: known allergy to mycophenolatmofetil, neutropenia, severe active gastrointestinal tract disease, Lesch-Nyhan syndrome or Kelley-Seegmiller syndrome, current intake of azathioprine
* cyclosporine: known allergy to cyclosporine, increased intracranial pressure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2007-03; Primary Completion 2011-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 3
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 6
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 9
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 12
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 15
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 18
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 21
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)
Progression of actinic keratosis or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors | at month 24
  Progression of actinic keratosis I and II to III or invasive squamous cell carcinoma (SCC) or incidence/reoccurrence of neoplastic skin tumors (namely SCC, basal cell carcinoma, keratoacanthoma, Bowen's disease, precancerous keratoses, actinic keratoses III)